CLINICAL TRIAL: NCT07007572
Title: Evaluation Of Marginal Bone Height Changes And Biting Force In Screw Retained Implant Prostheses Using Reinforced Resin Vs Monolithic Zirconium Used In Unilateral Distal Extension Cases
Brief Title: Evaluation Of Marginal Bone Height Changes And Biting Force In Screw Retained Implant Prostheses Using Reinforced Resin Vs Monolithic Zirconium
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Saleh Fayed, associate lecturer- prosthodontics department- faculty of dentistry, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 31-12-24
Record Dates: First submitted 2025-05-18; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Biting Forces; Bone; Change, Diabetic (Manifestation); Color Stability; Disorder of Soft Tissue; Prosthetic Complications; Bacterial Overgrowth
Keywords: biting forces; Bacterial Adhesion; color stability; soft tissue response; prosthetic complication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients who receives a screw retained monolithic zirconia bridge (Active Comparator): Digitally-fabricated implant supported supra-structure fabricated from monolithic zirconia
  Interventions: Combination Product: Digitally-fabricated implant supported supra-structure fabricated from reinforced resin
- patients who receives a screw retained resin reinforced bridge (Experimental): Digitally-fabricated implant supported supra-structure fabricated from reinforced resin
  Interventions: Combination Product: Digitally-fabricated implant supported supra-structure fabricated from monolithic zirconia

INTERVENTIONS:
Combination Product: Digitally-fabricated implant supported supra-structure fabricated from reinforced resin — A comprehensive clinical examination with an understanding of patients' chief complaints and needs will be carried out. For each patient, two implants will be placed in the edentulous area, and the patient will receive a screw-retained bridge supported by both implants made of milled monolithic zirconia (Dental Direkt Zirconia, Germany). After 6 months, the zirconia restoration will be replaced with a milled resin-reinforced composite (Nanoska G Plus, USA), allowing the same patient to use the new restoration for another 6 months. Randomization will be performed to determine the sequence of bridge material for each participant. Accordingly, the two restorations will be sequentially delivered to each participant with no gap (wash-up period) between them. Consent will be signed by the selected participants after explaining the detailed information of the trial.
  Arms: patients who receives a screw retained monolithic zirconia bridge
Combination Product: Digitally-fabricated implant supported supra-structure fabricated from monolithic zirconia — Digitally-fabricated implant supported supra-structure fabricated from monolithic zirconia
  Arms: patients who receives a screw retained resin reinforced bridge

SUMMARY:
This studies aims to compare the behavior of recently introduced resin reinforces compared to monolithic zirconia

DETAILED DESCRIPTION:
The clinical success of implant-supported prostheses is significantly influenced by the material used, as it directly affects both prosthetic longevity and patient satisfaction. Monolithic zirconia, despite its widespread popularity, presents notable clinical challenges. Its excessive rigidity often leads to mechanical failures such as chipping, fractures, and increased wear of the opposing dentition. Moreover, zirconia's limited ability to absorb and dissipate occlusal forces can result in elevated stresses on implant components, contributing to screw loosening or fractures and necessitating frequent maintenance interventions. These complications not only escalate the overall cost of care but also negatively impact patient outcomes, leading to discomfort, inconvenience, and dissatisfaction. Consequently, there is a pressing need to explore alternative restorative materials that maintain strength and esthetic appeal while mitigating these clinical issues. Biomimetic reinforced resin composites, engineered to emulate the mechanical behavior of natural tooth structures, offer a promising solution. By more effectively absorbing and distributing occlusal forces, these materials may reduce stress on both prostheses and surrounding tissues. If clinically validated, biomimetic resins could lead to fewer mechanical complications, improved bone preservation, and enhanced overall durability of implant-supported prostheses. The clinical implications of adopting biomimetic reinforced resin are substantial; a material that reduces the frequency of repairs and replacements compared to monolithic zirconia would mark a significant advancement in prosthetic dentistry, offering clinicians a superior restorative option and improving patient satisfaction through more stable, long-term outcomes.

To investigate this, mandibular Class II partially edentulous patients will be recruited from the outpatient clinic at the Department of Prosthodontics, Cairo University, based on specific inclusion criteria. After obtaining informed consent and conducting a comprehensive clinical examination, each patient will receive two implants in the edentulous area, restored initially with a screw-retained bridge made of milled monolithic zirconia. After six months, the zirconia bridge will be replaced with a milled resin-reinforced composite bridge. The sequence of material placement will be randomized for each participant, ensuring that each patient uses both materials sequentially without a washout period.

Intraoral scans and digital bite registrations will be performed, and prostheses will be designed using CAD software. Fabrication will follow standardized milling techniques for both zirconia and resin-reinforced composite materials. Bone levels around the implants will be evaluated using long cone parallel periapical radiographs, with measurements recorded at 0 and 6 months during each material phase. This approach allows for direct comparison of the two materials' effects on peri-implant bone health.

Biting forces will also be assessed using an occlusal force meter. A reference bite force will be measured on the intact side, followed by measurements on the intervention side after the placement of each restorative material. Each measurement will be repeated five times and averaged to ensure accuracy. All data regarding bone levels and biting forces will be recorded, tabulated, and statistically analyzed in the presence of an outcome assessor during clinical visits. Through this study design, it will be possible to evaluate the mechanical and biological performance of monolithic zirconia versus biomimetic reinforced resin composites in implant-supported prostheses.

ELIGIBILITY:
Inclusion Criteria:

* Mandibular Class II, partially edentulous patients that enables measuring the marginal bone height changes and values of biting forces intra-orally.
* Fully dentulous edentulous opposing Maxillary arch.
* Patients with normal class I jaw relationship.
* Patients that require fixed restorations for functional and esthetic reasons
* Age range (30-60 years).
* Cooperative patients those are willing to attend all follow-up periods.
* Patients with healthy attached mucosa of appropriate thickness free from any inflammation.
* Patients with healthy bone of appropriate thickness, width and height free from any inflammation.
* Patients without any medical conditions that contraindicates implant placement.

Exclusion Criteria:

* Patients with Parkinson's disease
* Patients with xerostomia.
* Patients with a history of allergy to resins and/ or zirconia.
* Patients with a medical systematic condition that contraindicate implant placement.
* Patients smoking more than 10 cigarettes per day.
* Patients with pathological changes of residual ridges as recurrent or persistent ulcers, osteomyelitis and infections.
* Patients with large irregular bony exostosis.
* Patients with medical or psychological conditions as physical disability or mental retardation that hinder cooperation in the follow up visits and answering the questionnaires.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of the Bone height changes (bone level) | 6 months for each arm
  Change in marginal bone height (in millimeters) measured using long cone parallel peri-apical radiographs at baseline and 6 months for each prosthetic material phase (monolithic zirconia and resin-reinforced). Radiographs will be taken at four time points:
  Start of phase 1 (zirconia, baseline)
  End of phase 1 (zirconia, 6 months)
  Start of phase 2 (resin-reinforced, baseline)
  End of phase 2 (resin-reinforced, 6 months)
  Bone level will be assessed on the mesial and distal surfaces of each implant using a standardized radiographic protocol.

SECONDARY OUTCOMES:
Average Maximum Biting Force | 6 months for each arm
  Average maximum static biting force (in Newtons) recorded using an occlusal force meter. For each prosthetic material phase (monolithic zirconia and resin-reinforced), patients will bite on the sensor five times per side. The average value from the intervention side (restored side) will be compared with that of the intact side. Measurements will be taken after prosthetic delivery for both phases and compared using statistical analysis to assess relative performance.
  Time Points:
  After placement of zirconia prosthesis
  After placement of resin-reinforced prosthesis
  Tool Used:
  Occlusal force meter with digital sensor, positioned on molars of both the intact and intervention sides.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
At this time, no final decision has been made regarding the sharing of individual participant data (IPD). The decision will depend on factors such as participant consent, institutional policies, data privacy considerations, and the potential for future collaborative research. If data sharing is approved, it will comply with all applicable ethical and legal standards.

REFERENCES:
- [Result] Roh, K.-W. et al. (2019) 'A prospective clinical of lithium disilicate pressed zirconia and monolithic zirconia in posterior implant-supported prostheses: A 24-month follow-up', The Journal of Korean Academy of Prosthodontics, 57(2), p. 134. doi: 10.4047/jkap.2019.57.2.134.
- [Result] Nitschke I, Moede C, Hopfenmuller W, Sobotta BAJ, Koenig A, Jockusch J. Validation of a New Measuring Instrument for the Assessment of Bite Force. Diagnostics (Basel). 2023 Nov 21;13(23):3498. doi: 10.3390/diagnostics13233498. PMID 38066739
- [Result] Liu, Y., Wang, S. and Chen, J. (2023) 'Challenges of monolithic zirconia in implant prosthodontics: Biting forces and maintenance considerations', Journal of Prosthetic Dentistry, 132(1), pp. 75-82. Available at: https://www.journals.elsevier.com/the-journal- of-prosthetic-dentistry.
- [Result] Lee, K. H., Patel, M. A. and Smith, A. D. (2023) 'Enhancing function and esthetics in partial edentulism: The role of biomimetic materials', Journal of Prosthetic Dentistry, 130(2), pp. 150-158. Available at: https://www.journals.elsevier.com/the-journal-of-prosthetic- dentistry.
- [Result] Gomez, P. H. et al. (2023) 'Advances in resin composites: A review of biomimetic approaches in prosthetic dentistry', Journal of Prosthetic Dentistry. Available at: https://www.journals.elsevier.com/the-journal-of-prosthetic-dentistry.
- [Result] Ahmed, N., Patel, A. and Zhang, X. (2024) 'Prosthetic Rehabilitation of Edentulous Patients: A Systematic Review of Complications and Management', International Journal of Prosthodontics, 37(2), pp. 214-223. doi: 10.11607/ijp.7698.

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2024-11-23): https://cdn.clinicaltrials.gov/large-docs/72/NCT07007572/Prot_ICF_000.pdf